CLINICAL TRIAL: NCT04921956
Title: Concizumab Compassionate Use Programme for Patients With Congenital Haemophilia
Brief Title: Compassionate Use of Concizumab if You Have Haemophilia
Status: Available | Type: Expanded Access
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7415-4807
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Congenital Haemophilia
MeSH Terms: interventions — concizumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Concizumab — Injected under the skin (subcutaneous, sc) once daily, individual dose adjustment.

SUMMARY:
The compassionate use programme will give participants concizumab for free, even though it is not yet approved by health authorities. This is because participants need this medicine to treat their haemophilia properly. The programme will check that participants are safe and that the medicine works for them. The programme may last for years. Participants will take one injection under their skin every day. Participants will have 4-5 visits with the study doctor for the first half year. After that they will have 1 visit every half year. At all clinic visits participants will have blood samples taken. Participants will fill in a diary between the visits.

A patient is considered to have completed the programme when any of the following criteria occurred first: 1) when the patient is included in a clinical trial with concizumab or 2) up to 6 months after concizumab is commercially available in the patient's country and approved for the patient (The time span of 6 months should provide ample time for the patient to obtain concizumab commercially) or 3) the sponsor decides to discontinue concizumab clinical development for the patient's population.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any programme-related activities. Programme-related activities are any procedures that are carried out as part of the programme.
* Patients with congenital haemophilia:

  1. severe haemophilia A (coagulation factor VIII (FVIII) less than 1%) or moderate/severe haemophilia B (coagulation factor IX (FIX) less than or equal to 2%) without inhibitors or
  2. any haemophilia severity with documented history of inhibitors (more than or equal to 0.6 bethesda unit (BU)) who cannot be treated satisfactorily with authorised and marketed medicines (example: due to inhibitors or allergic reactions to factor-containing products, or due to poor venous access), and who are not able to enrol in clinical trials designed to support the development and registration of concizumab medicines (example: due to inhibitors or allergic reactions to factor-containing products, or due to poor venous access) as per investigator and Novo Nordisk assessment.
* The potential benefit for the individual patient justifies the potential risks of treatment.

Exclusion Criteria:

* Known or suspected hypersensitivity to investigational medicinal product or related products.
* Any condition (current or medical history), which in the investigator's or Novo Nordisk's opinion might jeopardise patient's safety or compliance with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (25):
- United States (23):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - University of California San Francisco UCSF, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Augusta University, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - Childrens Hospital of Chicago, Chicago, Illinois
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - Children's Hospital of Michigan, Detroit, Michigan
  - Southern Specialty Clinic, Flowood, Mississippi
  - Louisiana Ctr for Adv Med-LCAM, Madison, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Children's Nebraska, Omaha, Nebraska
  - ECU Sickle Cell Comp Clinic, Greenville, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - BI-LO Chrt Childn's Cancer Ctr, Greenville, South Carolina
  - Cook Children's Hospital-Hematology-Oncology, Fort Worth, Texas
  - Texas Children's Hospital_Houston, Houston, Texas
  - Univ TX Hlth Sci Ctr Houston, Houston, Texas
  - Virginia Commonwealth University_Richmond_1, Richmond, Virginia
- UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Pediatrics, Plovdiv, Bulgaria
- Koagulationsmottagningen, Solna, Sweden